CLINICAL TRIAL: NCT00587015
Title: A Phase I, Multicenter, Dose Escalation Study of CAT-8015 in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL)
Brief Title: A Phase I, Multicenter, Dose Escalation Study of CAT-8015 in Patients With Non-Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to a lack of IP supply and then terminated because they were combined into one new study with the new IP formulation.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-8015-1003
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): CAT-8015
  Interventions: Drug: CAT-8015

INTERVENTIONS:
Drug: CAT-8015 — The dose level of the initial cohort will be 5 μg/kg so cohorts will be dosed at 5, 10, 20, 30, 40, 50, 60…μg/kg until toxicity supervenes.

SUMMARY:
A dose-escalation study to estimate the maximum tolerated dose(MTD) of CAT-8015 that can be safely administered to a patient.

DETAILED DESCRIPTION:
To estimate the maximum tolerated dose (MTD), defined as the highest dose that can be safely administered to a patient, and to establish a safe dose, based on MTD, for subsequent clinical testing.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible to participate in the study:

* Confirmed diagnosis of B-cell non-Hodgkin's lymphoma
* Measurable disease
* Evidence of CD22-positive malignancy by the following criteria, > 30% of malignant cells from a disease site CD22+ by FACS analysis or, > 15% of malignant cells from a disease site must react with anti-CD22 by immunohistochemistry
* Disease characteristics: Patients with indolent subtypes of CD22+ B-cell non- Hodgkin's lymphoma, including, but not limited to mantle cell lymphoma, follicular lymphoma and Waldenström's macroglobulinemia, are eligible if stage III-IV. if stage III-IV. Patients must have failed at least two or more courses of prior standard chemotherapy and/or biologic therapy (e.g. Rituxan). Patients with progressive mantle cell lymphoma may be eligible if they have failed one prior standard therapeutic regimen.
* ECOG performance status of 0-2
* Patients with other cancers who meet eligibility criteria and have less than 5 years of disease free survival will be considered on a case-by-case basis
* Life expectancy of less than 6 months, as assessed by the principal investigator
* Must be able to understand and sign informed consent
* Must be at least 18 years old
* Female and male patients must agree to use an approved method of contraception during the study

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for participation in the study:

* History of allogeneic bone marrow transplant
* Documented and ongoing central nervous system involvement with their malignant disease (history of CNS involvement is not an exclusion criterion)
* Pregnant or breast-feeding females
* HIV positive serology (due to increased risk of severe infection and unknown interaction of CAT-8015 with antiretroviral drugs)
* Hepatitis B surface antigen positive
* Uncontrolled, symptomatic, intercurrent illness including but not limited to: infections requiring systemic antibiotics, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements
* Patients whose plasma contains either a significant level of antibody to CAT-8015 as measured by ELISA, or antibody that neutralizes the binding of CAT-8015 to CD22 as measured by a competition ELISA.

Hepatic function Serum transaminases (either ALT or AST) or bilirubin:

* ≥ Grade 2, unless bilirubin is due to Gilbert's disease

Renal function:

* serum creatinine clearance ≤ 60mL/min as estimated by Cockroft-Gault formula

Hematologic function:

* The ANC < 1000/cmm, or platelet count <50,000/cmm, if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy).
* A patient will not be excluded because of pancytopenia ≥ Grade 3, or erythropoietin dependence, if it is due to disease, based on the results of bone marrow studies
* Baseline coagulopathy greater than or equal to Grade 3 unless due to anticoagulant therapy.

Pulmonary function:

* Patients with < 50% of predicted forced expiratory volume (FEV1) or <50% of predicted diffusing capacity for carbon monoxide (DLCO), corrected for hemoglobin concentration and alveolar volume. Note: Patients with no prior history of pulmonary illness are not required to have PFTs. FEV1 will be assessed after bronchodilator therapy.

Recent prior therapy:

* Cytotoxic chemotherapy, corticosteroids (except stable doses of prednisone), whole body electron beam radiation therapy, hormonal, biologic or other standard or any investigational therapy of the malignancy for 3 weeks prior to entry into the trial
* Less than or equal to 1 month prior monoclonal antibody therapy (i.e. rituximab)
* Patients who are receiving or have received radiation therapy less than 3 weeks prior to study entry will be not be excluded providing the volume of bone marrow treated is less than 10% and also the patient has measurable disease outside the radiation port
* Any history of prior pseudomonas-exotoxin immunotoxin (PE) administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Assess safety, estimate MTD, characterize toxicity profile, study pharmacology and observe anti-tumor activity at the MTD. | Day 28

SECONDARY OUTCOMES:
Assess immunogenicity of CAT 8015 and potential biomarkers for therapeutic or toxicity responses. | Day 0-7; 0-14

CONTACTS AND LOCATIONS:
Overall Officials: Robert Leechleider, M.D., Study Director — MedImmune LLC
Locations (3):
- United States (2):
  - Tower Hematology Oncology Medical Group, Beverly Hills, California
  - NCI, National Institutes of Health, Bethesda, Maryland
- Kalinika Hemotologii Uniwersytetu Medycznego, Lodz, Poland